CLINICAL TRIAL: NCT01069887
Title: A Non-interventional Multicentre Prospective Registry to Monitor the Incidence of Invasive Fungal Infections and to Monitor the Diagnostic and Therapeutic Management of Suspected Fungal-related Febrile Episodes in Patients With Malignant Hemopathies or Subjected to Haematopoietic Cell Transplant for the Treatment of Onco-haematological Diseases (HEMA E-CHART REGISTRY)
Brief Title: A Prospective Registry for Febrile Events in Patients With Malignant Hemopathies or Subjected to Haematopoietic Stem Cell Transplant
Acronym: HEMA E-CHART
Status: Completed | Type: Observational
Sponsor: Catholic University of the Sacred Heart (Other)
Collaborators: Pagano L, Aversa F, Locatelli F, Nosari A,Rossi G, Viale P (Unknown)
Other Study IDs: 578/06
Record Dates: First submitted 2010-02-16; First posted 2010-02-17 (Estimated); Last update posted 2010-02-24 (Estimated); Status verified 2009-04

CONDITIONS: Hematological Malignancies; Stem Cell Transplantation
Keywords: febrile events; invasive fungal infections; hematological patients
MeSH Terms: conditions — Hematologic Neoplasms; Invasive Fungal Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- adult with hematological malignancies
- pediatrics with hematological malignancies
- pediatrics receiving stem cell transplant
- adult receiving stem cell transplant

SUMMARY:
Hema e-chart is an electronic case record that can be changed in real time and is based on the chronological organisation of the infective events and the therapies prescribed. It allows the collection of all personal, epidemiological, diagnostic and therapeutic data pertaining to the patient, processing it and analysing the results.

Aims and objectives of the project

The aims of this registry are:

* To assess how many suspected fungal-related febrile episodes identify an infective fungal agent
* To have a clear view of the diagnostic and therapeutic actions in the management of onco-haematological patients with suspected fungal-related febrile episodes
* To assess the impact of anti-fungal therapy on the timing of chemotherapy and transplant planning
* Perform drug-epidemiology relationship analyses, observe toxicity and interactions with antifungal therapies by means of the creation of a national database of fungal infections in patients affected by malignant haemopathies

Design

* A multicentre, prospective registry for monitoring invasive fungal infections in onco-haematological patients
* Registration criteria: patients with newly diagnosed malignant haematological diseases (acute and chronic myeloid and lymphoid leukaemia, multiple myeloma, non-Hodgkin's and Hodgkin's lymphoma, aplastic anaemia, myelodysplastic syndromes), or patients who, as a result of onco-haematological pathologies, have undergone allogenic or autologous haematopoietic cell transplants, and have ongoing febrile episodes . The recording of consecutive febrile events is required
* Data collection for each individual patient will be performed according to the method shown in the enclosed flow chart. In the case of a new episode for an existing patient, said new episode will be recorded in the same case record as a new event. All collected data will be coded into the database
* Information relating to about 500 suspected fungal-related febrile events requiring antifungal therapy is expected to be collected from approximately 60 centres over the course of 18 months
* Data collection for each event may be performed following the provision of written informed consent, which will be obtained from each patient participating in this health survey
* The data collected will be handled and stored in full compliance with the Italian laws governing privacy
* Hema e-chart is a non-interventional registry

DETAILED DESCRIPTION:
Introduction Problems with infections in onco-haematological patients have assumed ever increasing importance over recent years, with relation to the development of management principles of the various clinical entities. Indeed, infections are primarily correlated with reduced immunocompetence (both cellular and humoral immunity) following both intensive chemotherapy and the use of immunosuppressant drugs during allotransplantation procedures. Furthermore, the common haematological disorders (i.e. acute or chronic myeloid and lymphoid leukaemia, lymphoma, myeloma etc) and the treatments required for such diseases contribute towards mediating and modulating the risk of infection. Among the various pathogens responsible for infections in onco-haematological patients, fungi still represent a problem for diagnosis and, despite the current therapeutic options, contribute significantly towards transplant-related mortality. The various candidaemias account for 30-40% of deaths, invasive aspergillosis for 50-60%, and 75% of deaths are accounted for by infections caused by zygomycetes.

Fungal agents include both the yeasts (e.g. Candida) and the moulds (e.g. Aspergillus, Zygomycetes); however over recent years, a different epidemiological trend has been observed between the aforementioned macro-categories of etiological agents: while there has been a progressive reduction in the epidemiological and clinical burden caused by Candida spp infections, the opposite trend has been observed for those caused by moulds, Aspergillus spp. and so on. Nevertheless, all clinicians are well aware of this epidemiological development the variables associated with risk and the real incidence of fungal infections in patients with malignant haemopathies and/or subjected to transplant are not entirely known. A recent multicentre retrospective study by the GIMEMA group assessed mould infections in patients with malignant haemopathies over a 10 year period. This study showed that 6-7% of patients with acute leukaemia can develop a mould infection during one of the various stages of the disease (onset of remission, relapse, rescue therapy, etc). Despite the undoubted use of this data as a first assessment of the magnitude of the problem, a more thorough epidemiological investigation appears in need, above all within the context of being able to plan the correct decisional procedure in relation to treatment, independently from the documentation of the infection. Secondly, an analysis of the different diagnostic approaches of the individual specialists, in terms of disease definitions and diagnostic work-up just as with their therapeutic choices, can contribute towards overcoming the high level of managerial empiricism still widespread within this medical sector.

The information which can be gathered from a study of this nature can prove useful for deducing the correct diagnostic approach and a suitable therapeutic decision, in day to day clinical practice. Hence, an integrated, computerised system, capable of recording the various different aspects, can certainly be of help to the haematology specialist.

Aims and objectives of the project

The aims of this registry are:

1. to assess how many suspected fungal-related febrile episodes identify an infective fungal agent.
2. to have a clear view of the diagnostic and therapeutic actions in the management of onco-haematological patients with suspected fungal-related febrile episodes.
3. to assess the impact of anti-fungal therapy on the timing of chemotherapy and transplant planning
4. perform drug-epidemiology relationship analyses, observe toxicity and interactions with antifungal therapies by means of the creation of a national database of fungal infections in patients affected by malignant haemopathies

Design

* A multicentre, prospective registry for monitoring invasive fungal infections in onco-haematological patients
* Registration criteria: patients with newly diagnosed malignant haematological diseases (acute and chronic myeloid and lymphoid leukaemia, multiple myeloma, non-Hodgkin's and Hodgkin's lymphoma, aplastic anaemia, myelodysplastic syndromes), or patients who, as a result of onco-haematological pathologies, have undergone allogenic or autologous haematopoietic cell transplants, and have ongoing febrile episodes . The recording of consecutive febrile events is required.
* Data collection for each individual patient will be performed according to the method shown in the enclosed flow chart. In the case of a new episode for an existing patient, said new episode will be recorded in the same case record as a new event. All collected data will be coded into the database.
* Information relating to approximately 500 suspected fungal-related febrile events requiring antifungal therapy is expected to be collected from approximately 60 centres over the course of 18 months.
* Data collection for each event may be performed following the provision of written informed consent, which will be obtained from each patient participating in this health survey.
* The data collected will be handled and stored in full compliance with the Italian laws governing privacy.
* Hema e-chart is a non-interventional registry.

The inclusion of patients in any given therapeutic strategy is not decided in advance, but falls within normal clinical practice, and the decision to prescribe any medication is entirely independent from that of including the patient in the health survey.

• Prior to its application, the plan will be submitted to the Ethics Committees of the various participating centres.

Data registration Hema e-chart is an electronic case record that can be changed in real time and is based on the chronological organisation of the infective events and the therapies prescribed. It allows the collection of all personal, epidemiological, diagnostic and therapeutic data pertaining to the patient, processing it and analysing the results. (see appendix).

This case record is located on a site with access controlled by user ID and Password Data registration will take place according to the method shown in the enclosed flow-chart

APPENDIX Hema e-chart Software The Hema e-chart software has been designed to be used in multiple specialised health centres. A configuration function allows automatic recognition of the centre to which the user submitting their access credentials belongs.

The data is structured according to the following general outline:

The patents basic personal data Description of the basic pathology Clinical parameters (neutrophils, temperature, etc) Disease type Type of treatment (1st line, 2nd line etc.) Drugs used Antibiotics Antivirals Antineoplastics Corticosteroids Immunomodulators Cytokines Renal function (calculated automatically as a function of creatinine levels) Hepatic function Diagnosis of fungal infection Chemical factors Microbiological factors Invasive tests Name of the fungal agent identified Site of infection Antifungal prophylaxis Antifungal agent selected Dosage Mode of administration Antifungal therapy Antifungal agent selected Dosage Mode of administration Outcome Outcome of the treatment

* Complete response (complete resolution of signs and symptoms, normalisation of any instrumental and/or mycological tests)
* Partial response (significant clinical improvement in both signs and symptoms and in any instrumental and/or mycological tests).

Physician's evaluation of the treatment Investigators comments Tolerability of the antifungal therapy Safety of the antifungal therapy Monitoring of any drug interactions

The Hema e-chart structure allows all the data contained in the case record to be altered and saved up to three times per day, while maintaining a complete history of all changes made. This way it is possible to follow the patient's progress, the treatments performed, the clinical tests requested, in detail, and then be able to assess any correlations existing between the actions undertaken and the effects obtained.

For this reason, the software is supplied with various graphical tools for easier evaluation of the data.

The same patient may be recorded several times in the study, if they incur several febrile events within the time period. Data registration allows use of the same personal details so as to aid consultation of the data.

ELIGIBILITY:
Inclusion Criteria:

* patients with newly diagnosed malignant haematological diseases (acute and chronic myeloid and lymphoid leukaemia, multiple myeloma, non-Hodgkin's and Hodgkin's lymphoma, aplastic anaemia, myelodysplastic syndromes), or patients who, as a result of onco-haematological pathologies, have undergone allogenic or autologous haematopoietic cell transplants, and have ongoing febrile episodes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with newly diagnosed malignant haematological diseases (acute and chronic myeloid and lymphoid leukaemia, multiple myeloma, non-Hodgkin's and Hodgkin's lymphoma, aplastic anaemia, myelodysplastic syndromes), or patients who, as a result of onco-haematological pathologies, have undergone allogenic or autologous haematopoietic cell transplants, and have ongoing febrile episodes
Sampling Method: Probability Sample
Enrollment: 3000 (Actual)
Dates: Start 2007-03; Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
number of febrile events | 3 times/week

SECONDARY OUTCOMES:
incidence of invasive fungal infections

CONTACTS AND LOCATIONS:
Locations (1):
- Hematology Institute - Catholic University, Rome, RM, Italy

REFERENCES:
- [Background] Pagano L, Girmenia C, Mele L, Ricci P, Tosti ME, Nosari A, Buelli M, Picardi M, Allione B, Corvatta L, D'Antonio D, Montillo M, Melillo L, Chierichini A, Cenacchi A, Tonso A, Cudillo L, Candoni A, Savignano C, Bonini A, Martino P, Del Favero A; GIMEMA Infection Program; Gruppo Italiano Malattie Ematologiche dell'Adulto. Infections caused by filamentous fungi in patients with hematologic malignancies. A report of 391 cases by GIMEMA Infection Program. Haematologica. 2001 Aug;86(8):862-70. PMID 11522544
- [Background] Muhlemann K, Wenger C, Zenhausern R, Tauber MG. Risk factors for invasive aspergillosis in neutropenic patients with hematologic malignancies. Leukemia. 2005 Apr;19(4):545-50. doi: 10.1038/sj.leu.2403674. PMID 15729382
- [Background] Martino R, Lopez R, Sureda A, Brunet S, Domingo-Albos A. Risk of reactivation of a recent invasive fungal infection in patients with hematological malignancies undergoing further intensive chemo-radiotherapy. A single-center experience and review of the literature. Haematologica. 1997 May-Jun;82(3):297-304. PMID 9234575
- [Result] Pagano L, Caira M, Nosari A, Viale P, Rossi G, Aversa F; Italian Hema e-Chart Group. Continuous surveillance of invasive fungal infection: a realistic goal for the near future. Clin Infect Dis. 2009 Jun 15;48(12):1801; author reply 1801-3. doi: 10.1086/599229. No abstract available. PMID 19473094
- [Derived] Pagano L, Caira M, Nosari A, Cattaneo C, Fanci R, Bonini A, Vianelli N, Garzia MG, Mancinelli M, Tosti ME, Tumbarello M, Viale P, Aversa F, Rossi G; HEMA e-Chart Group. The use and efficacy of empirical versus pre-emptive therapy in the management of fungal infections: the HEMA e-Chart Project. Haematologica. 2011 Sep;96(9):1366-70. doi: 10.3324/haematol.2011.042598. Epub 2011 May 12. PMID 21565903